CLINICAL TRIAL: NCT04538521
Title: NiaMIT (NiaMIT_0001) Continuation for Early-stage Mitochondrial Myopathy Patients to Investigate the Effect of Niacin Supplementation on Systemic Nicotinamide Adenine Dinucleotide (NAD+) Metabolism, Physiology and Muscle Performance
Brief Title: NiaMIT Continuation With Early-stage Mitochondrial Myopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other); Institute for Molecular Medicine (Other)
Responsible Party: Principal Investigator, Anu Wartiovaara, Academy Professor, Professor of Clinical Molecular Medicine; Chief Physician, University of Helsinki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NiaMIT_002
Record Dates: First submitted 2020-08-29; First posted 2020-09-04 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Mitochondrial Myopathies
Keywords: Vitamin B3; Niacin; Nicotinic acid; Mitochondrial myopathy; Mitochondria; Muscle; Muscle strength; Nicotinamide adenine dinucleotide; NAD+; NAD+ precursor; NAD-booster
MeSH Terms: conditions — Mitochondrial Myopathies | interventions — Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Niacin in early-stage mitochondrial myopathy patients (Experimental): The arm includes mitochondrial myopathy patients supplemented with niacin.
  Interventions: Dietary Supplement: Niacin

INTERVENTIONS:
Dietary Supplement: Niacin — The dose for a slow-released form of niacin will be 500-1000 mg/day. The daily niacin dose, 250 mg/day, is gradually escalated by 250 mg/month so that the full dose is reached after 2 months. The intervention time with the full niacin dose is 8 months and subsequently total intervention time 10 months.
  Other Names: Nicotinic acid

SUMMARY:
The most frequent form of adult-onset mitochondrial disorders is mitochondrial myopathy, often manifesting with progressive external ophthalmoplegia (PEO), progressive muscle weakness and exercise intolerance. Mitochondrial myopathy is often caused by single heteroplasmic mitochondrial DNA (mtDNA) deletions or multiple mtDNA deletions, the former being sporadic and latter caused by mutations in nuclear-encoded proteins of mtDNA maintenance. Currently, no curative treatment exists for this disease. However, an NAD+ precursor vitamin B3 has been demonstrated to give power to diseased mitochondria in animal studies by increasing intracellular levels of NAD+, the important cofactor required for the cellular energy metabolism. Vitamin B3 exists in several forms: nicotinic acid (niacin), nicotinamide, and nicotinamide riboside. Nicotinamide riboside has been shown to prevent and improve disease symptoms in several mouse models of mitochondrial myopathy. In addition, the investigators have previously observed that treatment with another form of vitamin B3, niacin, improved NAD+ deficiency and muscle performance in mitochondrial myopathy patients.

In this study, the form of vitamin B3, niacin, is used to activate dysfunctional mitochondria and to rescue signs of mitochondrial myopathy in early-stage patients. Of the vitamin B3 forms, niacin, is employed, because it has been used in large doses to treat hypercholesterolemia patients, and has a proven safety record in humans. Phenotypically similar mitochondrial myopathy patients are studied, as the investigator's previous expertise indicates that similar presenting phenotypes predict uniform physiological and clinical responses to interventions, despite varying genetic backgrounds. Patients with mitochondrial myopathy, typically harboring a sporadic single mtDNA deletion or a mutation in nuclear mtDNA maintenance gene causing multiple mtDNA deletions, are recruited. In addition, data from healthy controls from the primary NiaMIT study (ClinicalTrials.gov Identifier: NCT03973203) are utilized to analyse the collected data. Clinical examinations and collection of muscle biopsies are performed at the time points 0 and 10 months. Fasting blood samples are collected every second week until 1.5 months, every fourth week until 4 months and thereafter every six weeks until the end of the study. The effects of niacin on disease markers, muscle mitochondrial biogenesis, muscle strength and the metabolism of the whole body are studied in patients and healthy controls.

The hypothesis is that an NAD+ precursor, niacin, will increase intracellular NAD+ levels, improve mitochondrial biogenesis and alleviate the symptoms of mitochondrial myopathy already in early stages of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Early-stage, genetically diagnosed mitochondrial myopathy, with no major other symptoms or manifestations, caused by single or multiple deletions of mtDNA
2. Agreed to avoid vitamin supplementation or nutritional products with vitamin B3 forms 14 days prior to the enrollment and during the study
3. Written, informed consent to participate in the study

Exclusion Criteria:

1. Inability to follow study protocol
2. Pregnancy or breast-feeding at any time of the trial
3. Malignancy that requires continuous treatment
4. Unstable heart disease
5. Severe kidney disease requiring treatment
6. Severe encephalopathy
7. Regular usage of intoxicants

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
NAD+ and related metabolite levels in blood and muscle | Baseline, 4 months and 10 months
  Change in concentrations of NAD+ and related metabolites such as: nicotinamide adenine dinucleotide phosphate, nicotinic acid adenine dinucleotide, nicotinamide, and nicotinamide mononucleotide measured using a quantitative colorimetric assay.

SECONDARY OUTCOMES:
Number of diseased muscle fibers | Baseline and 10 months
  Change in number of abnormal muscle fibers (frozen sections, in situ histochemical activity analysis of cytochrome c oxidase negative / succinate-dehydrogenase positive muscle fibers; and immunohistochemistry of complex I negative muscle fibers
Mitochondrial biogenesis | Baseline and 10 months
  Change in mitochondria immunohistochemical staining intensity
Muscle mitochondrial oxidative capacity | Baseline and 10 months
  Change in muscle histochemical activity of mitochondrial cytochrome c oxidase
Muscle and blood metabolomic profiles | Baseline and 10 months
  Change in muscle or serum/plasma metabolite concentrations measured with mass spectrometry
Core muscle strength | Baseline and 10 months
  Change in core muscle strength measured by static and dynamic back and abdominal strength tests (number of repeats)
Circulating levels of disease biomarkers, fibroblast growth factor 21 (FGF21) and growth/differentiation factor 15 (GDF15) | Baseline and 10 months
  Change in circulating FGF21 and GDF15 concentrations measured using ELISA kits
Muscle mitochondrial DNA deletions | Baseline and 10 months
  Change in muscle mtDNA deletion load detected using polymerase chain reaction amplification
Muscle transcriptomic profile | Baseline and 10 months
  Change in muscle gene expression determined using RNA sequencing approach

OTHER OUTCOMES:
Body weight | Baseline and 10 months
  Change in body weight
Body composition | Baseline and 10 months
  Change in fat mass and fat free mass measured with bioimpedance
Ectopic lipid accumulation, i.e. liver and muscle lipid content | Baseline and 10 months
  Change in liver and muscle fat content measured with proton magnetic resonance spectroscopy
Circulating lipid profiles | Baseline, 4 months and 10 months
  Change in circulating HDL, LDL and triglyceride concentrations measured using standard photometric enzymatic assay

CONTACTS AND LOCATIONS:
Overall Officials: Anu Suomalainen Wartiovaara, MD, PhD, Principal Investigator — Research Program Unit, University of Helsinki, Helsinki, Finland
Locations (1):
- University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suomalainen A, Battersby BJ. Mitochondrial diseases: the contribution of organelle stress responses to pathology. Nat Rev Mol Cell Biol. 2018 Feb;19(2):77-92. doi: 10.1038/nrm.2017.66. Epub 2017 Aug 9. PMID 28792006
- [Background] Ylikallio E, Suomalainen A. Mechanisms of mitochondrial diseases. Ann Med. 2012 Feb;44(1):41-59. doi: 10.3109/07853890.2011.598547. Epub 2011 Aug 2. PMID 21806499
- [Background] Rajman L, Chwalek K, Sinclair DA. Therapeutic Potential of NAD-Boosting Molecules: The In Vivo Evidence. Cell Metab. 2018 Mar 6;27(3):529-547. doi: 10.1016/j.cmet.2018.02.011. PMID 29514064
- [Background] Khan NA, Auranen M, Paetau I, Pirinen E, Euro L, Forsstrom S, Pasila L, Velagapudi V, Carroll CJ, Auwerx J, Suomalainen A. Effective treatment of mitochondrial myopathy by nicotinamide riboside, a vitamin B3. EMBO Mol Med. 2014 Jun;6(6):721-31. doi: 10.1002/emmm.201403943. PMID 24711540
- [Background] Cerutti R, Pirinen E, Lamperti C, Marchet S, Sauve AA, Li W, Leoni V, Schon EA, Dantzer F, Auwerx J, Viscomi C, Zeviani M. NAD(+)-dependent activation of Sirt1 corrects the phenotype in a mouse model of mitochondrial disease. Cell Metab. 2014 Jun 3;19(6):1042-9. doi: 10.1016/j.cmet.2014.04.001. Epub 2014 May 8. PMID 24814483
- [Background] Vosper H. Niacin: a re-emerging pharmaceutical for the treatment of dyslipidaemia. Br J Pharmacol. 2009 Sep;158(2):429-41. doi: 10.1111/j.1476-5381.2009.00349.x. Epub 2009 Jul 20. PMID 19627285
- [Background] Guyton JR, Bays HE. Safety considerations with niacin therapy. Am J Cardiol. 2007 Mar 19;99(6A):22C-31C. doi: 10.1016/j.amjcard.2006.11.018. Epub 2006 Nov 28. PMID 17368274
- [Background] Ahola S, Auranen M, Isohanni P, Niemisalo S, Urho N, Buzkova J, Velagapudi V, Lundbom N, Hakkarainen A, Muurinen T, Piirila P, Pietilainen KH, Suomalainen A. Modified Atkins diet induces subacute selective ragged-red-fiber lysis in mitochondrial myopathy patients. EMBO Mol Med. 2016 Nov 2;8(11):1234-1247. doi: 10.15252/emmm.201606592. Print 2016 Nov. PMID 27647878
- [Background] Suomalainen A, Elo JM, Pietilainen KH, Hakonen AH, Sevastianova K, Korpela M, Isohanni P, Marjavaara SK, Tyni T, Kiuru-Enari S, Pihko H, Darin N, Ounap K, Kluijtmans LA, Paetau A, Buzkova J, Bindoff LA, Annunen-Rasila J, Uusimaa J, Rissanen A, Yki-Jarvinen H, Hirano M, Tulinius M, Smeitink J, Tyynismaa H. FGF-21 as a biomarker for muscle-manifesting mitochondrial respiratory chain deficiencies: a diagnostic study. Lancet Neurol. 2011 Sep;10(9):806-18. doi: 10.1016/S1474-4422(11)70155-7. Epub 2011 Aug 3. PMID 21820356
- [Background] Nikkanen J, Forsstrom S, Euro L, Paetau I, Kohnz RA, Wang L, Chilov D, Viinamaki J, Roivainen A, Marjamaki P, Liljenback H, Ahola S, Buzkova J, Terzioglu M, Khan NA, Pirnes-Karhu S, Paetau A, Lonnqvist T, Sajantila A, Isohanni P, Tyynismaa H, Nomura DK, Battersby BJ, Velagapudi V, Carroll CJ, Suomalainen A. Mitochondrial DNA Replication Defects Disturb Cellular dNTP Pools and Remodel One-Carbon Metabolism. Cell Metab. 2016 Apr 12;23(4):635-48. doi: 10.1016/j.cmet.2016.01.019. Epub 2016 Feb 25. PMID 26924217
- [Background] Khan NA, Nikkanen J, Yatsuga S, Jackson C, Wang L, Pradhan S, Kivela R, Pessia A, Velagapudi V, Suomalainen A. mTORC1 Regulates Mitochondrial Integrated Stress Response and Mitochondrial Myopathy Progression. Cell Metab. 2017 Aug 1;26(2):419-428.e5. doi: 10.1016/j.cmet.2017.07.007. PMID 28768179
- [Background] Pirinen E, Auranen M, Khan NA, Brilhante V, Urho N, Pessia A, Hakkarainen A, Kuula J, Heinonen U, Schmidt MS, Haimilahti K, Piirila P, Lundbom N, Taskinen MR, Brenner C, Velagapudi V, Pietilainen KH, Suomalainen A. Niacin Cures Systemic NAD+ Deficiency and Improves Muscle Performance in Adult-Onset Mitochondrial Myopathy. Cell Metab. 2020 Jun 2;31(6):1078-1090.e5. doi: 10.1016/j.cmet.2020.04.008. Epub 2020 May 7. PMID 32386566